# Informed Consent Form (ICF)

Official Title:

Clinical Evaluation of Kinesio Taping Outcomes in Stage II Cellulite: A Pilot Randomised Controlled Trial

NCT Number:

NCTXXXXXXXX

**Document Date:** 

September 16, 2025

Sponsor/Collaborator:

Klaipėda State University of Applied Sciences (Klaipėdos valstybinė kolegija)

#### 1. Introduction

You are invited to take part in a research study. Before you decide, it is important that you understand why the research is being done and what it will involve. Please take time to read the following information carefully.

## 2. Purpose of the Study

The purpose of this study is to evaluate whether kinesio taping applied to the thighs and buttocks can improve skin structure and reduce stage II cellulite. This is a pilot randomised controlled trial.

#### 3. Procedures

If you agree to participate, you will be randomly assigned to one of two groups:

- Experimental group: You will receive kinesio taping applied once weekly for four weeks.
- Control group: You will not receive kinesio taping during the study period.

All participants will undergo baseline and follow-up assessments including body composition, thigh circumference, cellulite evaluation, ultrasound of skin structure, and skin moisture measurements.

#### 4. Duration

Your participation in the study will last approximately 8 weeks, including 4 weeks of intervention and a 4-week follow-up.

#### 5. Risks and Discomforts

Kinesio taping is considered safe and non-invasive. Possible minor risks include temporary skin redness, itching, or irritation where the tape is applied. If you experience any discomfort, you may request removal of the tape.

#### 6. Benefits

You may or may not personally benefit from participating in this study. The results may help researchers and health professionals learn more about non-invasive treatments for cellulite.

## 7. Confidentiality

All information collected about you during the study will be kept confidential. Your data will be coded and stored securely. Results will be reported in a way that does not identify you personally.

### 8. Voluntary Participation and Withdrawal

Your participation is voluntary. You may refuse to participate or withdraw at any time without giving a reason, and without any penalty or loss of benefits to which you are otherwise entitled.

## 9. Compensation and Costs

There is no financial compensation for participation in this study. Participation is free of charge.

#### 10. Contact Information

If you have questions about the study, please contact the research team at PILDAU Clinical Research Unit. If you have questions about your rights as a participant, please contact the Ethics Committee of Klaipėda State University of Applied Sciences.

#### 11. Consent Statement

I have read and understood the information provided above. I have had the opportunity to ask questions and received satisfactory answers. I voluntarily agree to participate in this study.

| Participant's Name: | _ |
|--------------------------|-------|
| Participant's Signature: | Date: |
| Researcher's Name: | - |
| Researcher's Signature | Data: |